CLINICAL TRIAL: NCT03007745
Title: Remote Ambulatory Management of Veterans With Sleep Apnea
Brief Title: Remote Diagnosis and Management of Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 12-409
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Results first posted 2025-04-29 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Sleep Apnea - Obstructive; Cost Effectiveness; Telemedicine
Keywords: Continuous positive airway pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- REVAMP (Experimental): Veterans randomized to this arm will have access to the Remote Veteran Apnea Management Platform (REVAMP) a personalized, interactive website that allows Veterans to be evaluated for OSA without travelling to the sleep center.
  Interventions: Device: autoadjusting continuous positive airway pressure
- In-person management (Active Comparator): Veterans randomized to this arm will receive standard in-person management of their sleep apnea in the sleep center.
  Interventions: Device: autoadjusting continuous positive airway pressure

INTERVENTIONS:
Device: autoadjusting continuous positive airway pressure — Participants in both arms who are diagnosed with obstructive sleep apnea will be treated with autoadjusting continuous positive airway pressure
  Other Names: APAP

SUMMARY:
Although obstructive sleep apnea, a breathing disorder during sleep, is prevalent and recognized as a major public health concern, most Veterans with this disorder are undiagnosed and therefore untreated. Access to sleep laboratories for testing is limited particularly for those Veterans living in rural areas and Veterans with disabilities that prevent travel to a sleep center. The goal of this study is to compare a web-based telehealth management strategy to in-person management. The telehealth pathway will enable Veterans to be diagnosed and treated without visiting a sleep center. The investigators believe that telehealth management will increase Veterans' access to this specialized care at a cost that is less than in-person delivery but with similar improvements in daytime function.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is estimated to be the third most common chronic disease in Veterans and is associated with an increased risk of hypertension, heart attacks, strokes, depression, and driving accidents. Current in-person management at a sleep center limits Veterans' access to care, prolongs patient wait times, and requires Veterans living in remote areas to travel long distances. This proposal will evaluate an innovative web-based clinical pathway to diagnose and manage Veterans with OSA. In Fiscal Year 13, the investigative team received a Veterans Health Administration (VHA) Innovation Award to create the Remote Veteran Apnea Management Portal (REVAMP), a personalized, interactive website that, when combined with other emerging telehealth technologies, is designed to improve access to care, reduce patient wait times, and allow Veterans to receive care without travelling to a sleep center. Veterans complete intake and follow-up questionnaires on the REVAMP website and perform an unattended home sleep test (HST) without in-person instructions. Sleep specialists review the findings with the patient during an initial phone clinic. REVAMP auto-populates the Veteran's questionnaire responses into templated progress notes that are exported to CPRS, the electronic medical record. Veterans diagnosed with OSA are treated with automatically adjusting positive airway pressure (APAP) units. These devices transmit data wirelessly to the website where treatment use and its effectiveness can be monitored by both Veterans and practitioners, thereby promoting patient self-management and productive patient-practitioner interactions.

The investigators' proposed prospective, randomized intervention will compare the clinical and cost-effectiveness of REVAMP management of Veterans with OSA to in-person care. Aim 1 will determine if management with REVAMP is clinically non-inferior to in-person care in terms of improvement in functional outcomes and APAP adherence. Non-inferiority of clinical effectiveness following 3 months of APAP treatment will be expressed in terms of improvement in the score of the Functional Outcomes of Sleep Questionnaire (FOSQ-10), the investigators' primary outcome measure. Adherence to APAP will be objectively monitored by wireless transmission of data from the participant's home unit. In Aim 2, patient preference, medical service use and cost will be collected every 3 months for the entire observation period to compare cost effectiveness of the two managements. Preference will be assessed by the Short Form-6D (SF 6D), and the EuroQol-5D (EQ-5D). Differences in the ratio of cost and quality-adjusted life years saved by REVAMP compared to in-person management will test the hypothesis that REVAMP management will have lower cost and equivalent outcomes. The results of Aims 1 and 2 will provide evidence to support widespread dissemination of REVAMP. Formative evaluation in Aim 3 will use qualitative (targeted phone interviews) and quantitative measures (attrition, work alliance, and patient satisfaction) to inform clinicians, administrators and other stakeholders how to implement this innovative chronic disease pathway.

Aim 1 (primary). To compare functional outcomes following 3 months of APAP treatment in Veterans with OSA randomized to REVAMP versus in-person management. The primary outcome measure in this modified intent-to-treat analysis (i.e., subjects initiated on APAP with at least one FOSQ follow-up score) will be the change from baseline in the FOSQ-10 score. Analysis will also compare the mean daily hours of APAP use in participants in the two groups initiated on APAP treatment.

Hypothesis 1a: Mean change in FOSQ-10 score among participants randomized to REVAMP management will be no more than one point less than that in participants receiving in-person management.

Hypothesis 1b: Mean daily hours of APAP use among participants receiving REVAMP management will be no more than 0.75 hour less than that in participants randomized to in-person management.

Aim 2 (secondary): To compare the differences in cost and quality-adjusted life years (QALY) between REVAMP management and in-person management. The perspective of the analysis will be that of the VA and the intention to treat analysis set will include all randomized participants.

Hypothesis 2a: Average total health-care delivery cost will be lower for participants receiving REVAMP compared to in-person management.

Hypothesis 2b: The 90% lower limit of cost per QALY ratio comparing in-person versus REVAMP manage-ment will be > $100,000 (i.e., the investigators will have 90% confidence that REVAMP is good value for the cost).

Aim 3 (exploratory): To conduct a mixed methods formative evaluation that will guide REVAMP's widespread implementation. Quantitative component: The investigators will track quantitative outcome measures across both groups including attrition, participant- and practitioner-rated therapeutic alliance (Working Alliance Inventory-Short Revised [WAI-SR]),9 and participant treatment satisfaction (Client Satisfaction Questionnaire [CSQ-8]).10 The investigators will compare the scores of the WAI-SR and CSQ-8 and attrition rates between treatment arms. Qualitative component: The investigators will explore participant- and practitioner-level perspectives, attitudes, and preferences regarding REVAMP versus in-person management, as well as barriers and facilitators to participation in either clinical pathway through phone interviews with participants from the two intervention groups, participants who withdraw from either intervention, and staff who provide care through REVAMP.

Our primary aim was to demonstrate that the efficacy of REVAMP management is not clinically inferior to in-person care. Efficacy was measured as the change in FOSQ-10 score from pretreatment to 3 months following initiation of APAP treatment. An increase of more than 1 point in mean FOSQ score is felt to indicate an important clinical difference. Based on previous studies, we assumed a common SD=2.80. Similar calculations were performed for the APAP adherence outcome based on a non-inferiority delta of -0.75 hr/day and assuming a SD=2.2. 114 participants/group were estimated to be required to achieve at least 85% power to reject the null hypothesis, i.e., find that the change in FOSQ score among patients receiving the telehealth-based management is > 1 point lower than that in participants assessed in-person and that APAP adherence among participants receiving the telehealth-based management is > 0.75 hours lower that that in participants assessed in-person.

ELIGIBILITY:
Inclusion Criteria:

Veterans must meet the following inclusion criteria prior to enrollment:

* Referral to one of the participating sleep centers for evaluation of suspected OSA
* Access in the home to the internet, e-mail, and phone on all days
* Fluent in English as assessed on the initial phone contact

Exclusion Criteria:

Veterans will be excluded from the study for the following reasons:

* Unable or unwilling to provide informed consent and complete required questionnaires
* Previous diagnosis of:

  * obstructive sleep apnea (OSA)
  * central sleep apnea (50% of apneas on diagnostic testing are central apneas)
  * Cheyne-Stokes breathing
  * obesity hypoventilation syndrome
  * narcolepsy
* Previous treatment with positive airway pressure, non-nasal surgery for OSA, or current use of supplemental oxygen
* A clinically unstable medical condition in the previous 2 months as defined by a new diagnosis, e.g.:

  * pneumonia
  * myocardial infarction
  * congestive heart failure
  * unstable angina
  * thyroid disease
  * depression or psychosis
  * ventricular arrhythmias
  * cirrhosis
  * surgery
  * recently diagnosed cancer
* Night shift workers in situations or occupations where they regularly experience jet lag, or have irregular work schedules by history over the last 3 months
* Women who are pregnant or women who are sexually active and of child-bearing age who are not using some form of contraceptive
* Unable to perform tests due to inability to communicate verbally, inability to read and write, and visual, hearing or cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel T. Kuna, MD, Principal Investigator — Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA
Locations (3):
- United States (3):
  - VA San Diego Healthcare System, San Diego, CA, San Diego, California
  - Atlanta VA Medical and Rehab Center, Decatur, GA, Decatur, Georgia
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, PA, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang YHA, Folmer RL, Shasha B, Shea JA, Sarmiento K, Stepnowsky CJ, Lim D, Pack A, Kuna ST. Barriers and facilitators to the implementation of a novel web-based sleep apnea management platform. Sleep. 2021 Apr 9;44(4):zsaa243. doi: 10.1093/sleep/zsaa243. PMID 33216916

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | REVAMP | In-person Management
Started | 218 | 217
Completed | 85 | 114
Not Completed | 133 | 103
Not completed — Sleep test negative for OSA | 53 | 49
Not completed — Physician Decision | 6 | 9
Not completed — Withdrawal by Subject | 38 | 16
Not completed — Lost to Follow-up | 19 | 25
Not completed — Unable to login to website | 17 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | REVAMP | In-person Management | Total
Number analyzed (Participants) | 218 | 217 | 435
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.25 (13.31) | 47.25 (13.31) | 46.76 (13.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 88
  Male | 174 | 173 | 347
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian | 3 | 4 | 7
  Asian | 15 | 10 | 25
  Native Hawaiian | 2 | 3 | 5
  Black/African American | 92 | 111 | 203
  White | 95 | 78 | 173
  Unknown | 11 | 11 | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 218 | 217 | 435
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — Body mass index is calculated as body weight (kg) divided by height squared (meters) Population: Missing data
  kg/m2
    number analyzed (Participants) | 215 | 207 | 422
    (all) | 32.53 (5.46) | 32.87 (5.99) | 32.70 (5.72)
Apnea-hypopnea index (AHI) [Mean (Standard Deviation); unit: number of events/hour] — Scores for adults are divided into three categories, which correspond to different levels of obstructive sleep apnea severity. The apnea-hypopnea index (AHI) range is from 0 to ~140. It is true there is no upper true maximum, but above 140 is extremely unlikely:
  Normal: An AHI between 0 and fewer than 5. Mild severity: An AHI of at least 5 events per hour, but fewer than 15. Moderate severity: An AHI of at least 15 events per hour, but fewer than 30. Severe severity: An AHI of at least 30 events per hour. Population: missing data
  number of events/hour
    number analyzed (Participants) | 167 | 175 | 342
    (all) | 18.54 (24.58) | 20.71 (20.68) | 19.65 (22.66)
Oxygen desaturation index [Mean (Standard Deviation); unit: index] — Oxygen desaturation index is the average number of oxygen desaturation events with a 4% or greater drop from baseline during the analysis portion of the sleep study. The index is reported as events/hour. The oxygen desaturation index range is from 0 to ~140. There is no true upper maximum, but above 140 is extremely unlikely: A value of 5 events/hr or greater is considered abnormal. Higher values represent worse results. Population: Missing data
  index
    number analyzed (Participants) | 167 | 171 | 338
    (all) | 15.56 (22.93) | 17.7 (21.22) | 16.60 (21.99)
Functional Outcome of Sleep Questionnaire-10 [Mean (Standard Deviation); unit: units on a scale] — FOSQ-10 score ranges between 5 and 20 units; there is not threshold for normality; a higher score indicates higher functional outcome. Population: missing data
  units on a scale
    number analyzed (Participants) | 141 | 188 | 329
    (all) | 12.51 (3.86) | 12.92 (3.69) | 12.75 (3.77)
Epworth Sleepiness Scale [Mean (Standard Deviation); unit: units on a scale] — The Epworth Sleepiness Scale score ranges from 0 to 24 units; a value less than 11 is considered within normal range; a value of 11 or greater is considered to indicate the presence of subjective daytime sleepiness. Population: missing data
  units on a scale
    number analyzed (Participants) | 141 | 184 | 325
    (all) | 12.07 (5.56) | 12.28 (5.70) | 12.19 (5.63)
Insomnia Severity Index [Mean (Standard Deviation); unit: units on a scale] — Insomnia Severity Index scores range from 0 to 28 units with higher values indicating greater severity. Scores less than 8 are considered in the normal range. Scores between 8 and 14 are considered subthreshold insomnia. Scores between 15 and 21 are considered clinical insomnia of moderate severity and scores between 22 and 28 are considered severe clinical insomnia. Population: missing data
  units on a scale
    number analyzed (Participants) | 141 | 182 | 323
    (all) | 17.13 (6.19) | 16.75 (6.78) | 16.92 (6.53)
Pittsburgh Sleep Quality Index [Mean (Standard Deviation); unit: units on a scale] — The Pittsburgh Sleep Quality Index (PSQI) global score has a range of 0-21; higher scores indicate worse sleep quality. A global score less than or equal to 5 is felt to distinguish good from poor sleepers. Population: missing data
  units on a scale
    number analyzed (Participants) | 141 | 170 | 311
    (all) | 13.52 (3.52) | 13.74 (3.52) | 13.63 (3.52)
Medical Outcomes Study Short Form 12 (physical) [Mean (Standard Deviation); unit: units on a scale] — Medical Outcomes Study Short Form (physical) score ranges from 0 to 100. A higher score indicates a higher level of health or functioning. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health. Population: missing data
  units on a scale
    number analyzed (Participants) | 133 | 177 | 310
    (all) | 24.68 (0.40) | 24.65 (0.39) | 24.66 (0.40)
Medical Outcomes Study Short Form (mental) [Mean (Standard Deviation); unit: units on a scale] — Medical Outcomes Study Short Form (mental) score ranges from 0 to 100. A higher score indicates a higher level of health or functioning. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health. Population: missing data
  units on a scale
    number analyzed (Participants) | 133 | 177 | 310
    (all) | 18.24 (0.78) | 18.39 (0.75) | 18.32 (0.77)
European Quality of Life Visual Analogue Scale (EurQol-5D VAS) [Mean (Standard Deviation); unit: units on a scale] — The European Quality of Life Visual Analogue Scale (EurQol-5D VAS) is a visual vertical graduated analogue scale (ranging from 1 to 100) on which the participant self-rates health status. The score is reported as the units on the scale. Higher scores indicate better health status. The EurQol-5D does not have a cut-off threshold to distinguish good versus poor health status. Population: missing data
  units on a scale
    number analyzed (Participants) | 126 | 183 | 309
    (all) | 67.42 (16.71) | 64.97 (18.88) | 65.97 (18.04)
Center for Epidemiologic Studies Depression questionnaire (CES-D) [Mean (Standard Deviation); unit: units on a scale] — Center for Epidemiologic Studies Depression questionnaire (CES-D) is a 20-item standard instrument devised using items from 5 validated depression scales. Likert-style responses for each symptom indicates how often in the past week the subject has experienced the symptom. Scores on the CES-DC range from 0 to 60, in which higher scores suggest a greater presence of depressive symptoms. A score of 15 or higher is interpreted to indicate a risk for depression. Population: Missing data
  units on a scale
    number analyzed (Participants) | 142 | 186 | 328
    (all) | 13.38 (7.59) | 12.66 (6.49) | 12.97 (6.99)

OUTCOME MEASURES:

1. Primary Outcome: Functional Outcome of Sleep Questionnaire - Short Form (FOSQ-10)
Description: FOSQ-10 score ranges between 5 and 20 units; there is not threshold for normality; a higher score indicates higher functional outcome.
  Outcome Measure: Change from baseline in Functional Outcome of Sleep Questionnaire - Short Form (FOSQ-10), a self-administered disease specific quality of life questionnaire, in participants initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data). A change in 1 unit is felt to indicate clinical significance.
Time Frame: 3 months
Population: in participants initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REVAMP | In-person Management
Number analyzed (Participants) | 47 | 91
score on a scale | 1.96 (3.08) | 1.73 (3.97)
Statistical Analysis 1: Comparison: REVAMP; Paired t-test comparing baseline and 3-month measures within group; Test type: Superiority; p < 0.0001, t-test, 2 sided — Unadjusted; Mean Difference (Final Values) = 1.96, Standard Deviation 3.08
Statistical Analysis 2: Comparison: In-person Management; Paired t-test comparing baseline and 3-month measures within group; Test type: Superiority; p < 0.0001, t-test, 2 sided; Unadjusted; Mean Difference (Final Values) = 1.73, Standard Deviation 3.97
Statistical Analysis 3: Comparison: REVAMP vs In-person Management; Adjusted differences in mean changes were estimated as site-total-sample-size weighted values controlling for treatment group differences in mean pre-treatment baseline values. ANCOVA model included main effects for type of study (home versus in-laboratory), site, and the pre-treatment baseline value of the outcome measure; Test type: Superiority; p = 0.9171, ANCOVA — Adjusted mean changes and adjusted differences in mean changes were estimated as site-total-sample-size weighted values controlling for treatment group differences in mean pre-treatment baseline values; Mean Difference (Final Values) = -0.06, Standard Error of Mean 0.61
Statistical Analysis 4: Comparison: REVAMP vs In-person Management; Test type: Non-Inferiority — We hypothesized that the lower bound of the non-inferiority analysis of FOSQ-10 would be greater than the a-priori threshold of -1.0; p > 0.05, ANCOVA — Adjusted group difference in mean change in FOSQ-10 score from baseline to Month 3, controlling for baseline FOSQ and site, was -0.06 ± 061 (SEM) (P = 0.917). The lower bound of the 95% noninferiority confidence interval was -1.08

2. Secondary Outcome: Epworth Sleepiness Scale (ESS)
Description: Epworth Sleepiness Scale score ranges from 0 to 24 units; a value less than 11 is considered within normal range; a value of 11 or greater is considered to indicate the presence of subjective daytime sleepiness.
  Outcome measure: Change from baseline in the Epworth Sleepiness Scale (ESS), a self-administered subjective measure of daytime sleepiness, in participants initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data). A score change of 2 units is felt to indicate clinical significance.
Time Frame: 3 months
Population: Subjects initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REVAMP | In-person Management
Number analyzed (Participants) | 48 | 91
score on a scale | -3.31 (4.86) | -3.51 (5.52)
Statistical Analysis 1: Comparison: REVAMP; Paired t-test comparing baseline and 3-month measures within group; Test type: Superiority; p < 0.0001, t-test, 2 sided — Subjects initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data) Paired t-test comparing baseline and 3-month measures within group; Mean Difference (Net) = -3.31, Standard Deviation 4.86
Statistical Analysis 2: Comparison: In-person Management; Subjects initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data) Paired t-test comparing baseline and 3-month measures within group; Test type: Superiority; p < 0.0001, t-test, 2 sided — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Net) = -3.51, Standard Deviation 5.52
Statistical Analysis 3: Comparison: REVAMP vs In-person Management; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.9251, ANCOVA; ANCOVA included main effects for group, site, and the pre-treatment baseline value of the outcome measure; Mean Difference (Final Values) = 0.08, Standard Error of Mean 0.85

3. Secondary Outcome: Heath Survey Short Form - 12 (SF-12) Physical Component
Description: Medical Outcomes Study Short Form (physical) score ranges from 0 to 100. A higher score indicates a higher level of health or functioning. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health. Outcome measure: Change from baseline in physical component of the Health Survey Short Form-12 (SF-12), a self administered quality of life questionnaire, in participants initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data).
Time Frame: 3 months
Population: Subjects initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REVAMP | In-person Management
Number analyzed (Participants) | 46 | 84
score on a scale | 0.04 (0.33) | -0.05 (0.39)
Statistical Analysis 1: Comparison: REVAMP; Within arm change from baseline to 3 month follow-up; Test type: Superiority — Paired t-test comparing change in score (3-month - baseline) within group; p = 0.4116, t-test, 2 sided; Subjects initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data); Mean Difference (Final Values) = 0.04, Standard Deviation 0.33
Statistical Analysis 2: Comparison: In-person Management; Paired t-test comparing change in score (3-month - baseline) within group; Test type: Superiority; p = 0.2201, t-test, 2 sided; Mean Difference (Net) = -0.05, Standard Deviation 0.39
Statistical Analysis 3: Comparison: REVAMP vs In-person Management; Adjusted differences in mean changes between groups from baseline to month 3 in participants initiated on CPAP (LOCF applied using 1-month data); Test type: Superiority; p = 0.1732, ANCOVA; ANCOVA included main effects for group, site, and the pre-treatment baseline value of the outcome measure; Mean Difference (Net) = 0.08, Standard Error of Mean 0.06

4. Secondary Outcome: Center for Epidemiological Studies Depression Questionnaire (CES-D)
Description: Center for Epidemiological Studies Depression Scale (CES-D) is a 20-item standard instrument devised using items from 5 validated depression scales. Likert-style responses for each symptom indicates how often in the past week the subject has experienced the symptom. Scores on the CES-DC range from 0 to 60, in which higher scores suggest a greater presence of depressive symptoms. A score of 15 or higher is interpreted to indicate a risk for depression.
  Outcome measure: Change from baseline in Center for Epidemiological Studies Depression questionnaire (CES-D), a self-administered assessment of depression, in participants initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data)
Time Frame: 3 months
Population: Subjects initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REVAMP | In-person Management
Number analyzed (Participants) | 45 | 91
score on a scale | -2.76 (4.73) | -2.38 (5.20)
Statistical Analysis 1: Comparison: REVAMP; Paired t-test comparing baseline and 3-month measures within group; Test type: Superiority; p < 0.0003, t-test, 2 sided; Unadjusted; Mean Difference (Final Values) = -2.76, Standard Deviation 4.73
Statistical Analysis 2: Comparison: In-person Management; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, t-test, 2 sided; Unadjusted; Mean Difference (Final Values) = -2.38, Standard Deviation 5.20
Statistical Analysis 3: Comparison: REVAMP vs In-person Management; Adjusted differences in mean changes were estimated as site-total-sample-size weighted values controlling for treatment group differences in mean pre-treatment baseline values. Subjects initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data); Test type: Superiority; p = 0.6730, ANCOVA; ANCOVA included main effects for group, site, and the pre-treatment baseline value of the outcome measure; Median Difference (Final Values) = -0.38, Standard Error of Mean 0.90

5. Secondary Outcome: Insomnia Severity Index (ISI)
Description: Insomnia Severity Index scores range from 0 to 28 units with higher values indicating greater severity. Scores less than 8 are considered in the normal range. Scores between 8 and 14 are considered subthreshold insomnia. Scores between 15 and 21 are considered clinical insomnia of moderate severity and scores between 22 and 28 are considered severe clinical insomnia.
  Outcome measure: Change from baseline of the Insomnia Severity Index (ISI), a aelf-administered assessment of insomnia, in participants initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data)
Time Frame: 3 months
Population: Change from baseline in subjects initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REVAMP | In-person Management
Number analyzed (Participants) | 47 | 89
score on a scale | -5.94 (6.17) | -5.60 (0.39)
Statistical Analysis 1: Comparison: REVAMP; Paired t-test comparing baseline and 3-month measures within group (LOCF applied using 1-month data); Test type: Superiority; p < 0.0001, t-test, 2 sided — Unadjusted; Paired t-test comparing baseline and 3-month measures within group (LOCF applied using 1-month data); Mean Difference (Net) = -5.94, Standard Deviation 6.17
Statistical Analysis 2: Comparison: In-person Management; Subjects initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data); Test type: Superiority — Paired t-test comparing baseline and 3-month measures within group (LOCF applied using 1-month data); p = 0.0001, t-test, 2 sided — Unadjusted; Mean Difference (Final Values) = -5.60, Standard Deviation 6.96
Statistical Analysis 3: Comparison: REVAMP vs In-person Management; Between group comparison of change in Insomnia Severity Index (ISI) at 3 months (LOCF applied using 1-month data); Test type: Superiority; p = 0.9903, ANCOVA — ANCOVA included main effects for group, site, and the pre-treatment baseline value of the outcome measure; Adjusted differences in mean changes estimated as site-total-sample-size weighted values controlling for group differences in mean baseline values; Mean Difference (Net) = 0.01, Standard Error of Mean 1.11

6. Secondary Outcome: Health Utilities Index (HUI)
Description: Health Utilities Index (HUI-2), a self-administered questionnaire on overall functional health, in participants initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data). HUI-2 classification system consists of 7 attributes including sensation, mobility, emotion, cognition, self-care, pain and fertility. HUI-2 utility values range from -0.03 to 1.00. A health utility value of 1.00 indicates perfect health while a score of 0.00 indicates death. To calculate a health utility score, health states for each response are converted using a look-up table and mathematical formula.
Time Frame: 3 months
Population: Veterans randomized to REVAMP vs In-person management. The reduced number of participants analyzed was due to missing data. In particular, many participants in the REVAMP arm failed to complete the on-line HUI questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REVAMP | In-person Management
Number analyzed (Participants) | 10 | 72
score on a scale | 0.7036 (0.2729) | 0.7165 (0.2127)

7. Secondary Outcome: EuroQol (EQ-5D) VAS
Description: EurQol-5D VAS is a visual vertical graduated analogue scale (ranging from 1 to 100) on which the participant self-rates health status. The score is reported as the units on the scale. Higher values represent a better health status. The EurQol-5D does not have a cut-off threshold to distinguish good versus poor health status.
  Outcome measure: Change from baseline in the EurQol-5D VAS score in participants initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REVAMP | In-person Management
Number analyzed (Participants) | 11 | 77
score on a scale | 68.82 (25.34) | 67.32 (20.85)

8. Secondary Outcome: Worker Alliance Inventory - Short Revised (WAI-SR)
Description: WAI-SR is the 12-item questionnaire to assess three key aspects of the therapeutic alliance: (a) agreement on the tasks of therapy, (b) agreement on the goals of therapy and (c) development of confidence, trust, comfort, and acceptance. Scores of each of the three key aspects range from 5 to 25 and the total WAI-SR score is the sum of the three subscored (maximum 75). Higher scores indicate greater alliance.
  Outcome measure: Assessment of participant-rated alliance with the practitioner in participants initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data)
Time Frame: 3 months
Population: Total client score in participants initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data) who completed the self-administered questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REVAMP | In-person Management
Number analyzed (Participants) | 8 | 74
score on a scale | 56.38 (19.32) | 64.68 (12.73)

9. Secondary Outcome: Client Satisfaction Questionnaire (CSQ-8)
Description: Client Satisfaction Questionnaire (CSQ-8) is an 8-item, self-administered structured survey used to assess level of satisfaction with care. Items are scored on a Likert scale from 1 (low satisfaction) to 4 (high satisfaction) with different descriptors for each response point. Total scores range from 8 to 32, with higher scores indicating greater satisfaction.
Time Frame: 3 months
Population: CSQ-8 score of participants initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REVAMP | In-person Management
Number analyzed (Participants) | 18 | 74
score on a scale | 19.44 (1.46) | 19.84 (2.03)
Statistical Analysis 1: Comparison: REVAMP vs In-person Management; Between group comparison of Client Satisfaction Questionnaire (CSQ-8) at 3 months (LOCF applied using 1-month data); Test type: Superiority; p > 0.05, t-test, 2 sided

10. Secondary Outcome: Adherence to Autoadjusting CPAP Treatment
Description: Objective assessment of adherence to CPAP treatment; average daily use over all days (hours)
Time Frame: 3 months
Population: Participants initiated on CPAP and receiving a 3-month follow-up (LOCF applied using 1-month data)
Measure: Mean (Standard Deviation); unit: hours per day
Arm/Group | REVAMP | In-person Management
Number analyzed (Participants) | 85 | 114
hours per day | 3.29 (2.65) | 2.91 (2.59)
Statistical Analysis 1: Comparison: REVAMP vs In-person Management; Test type: Non-Inferiority — The a-priori lower bound selected for the non-inferiority analysis of average daily CPAP use over 3 months was -0.75 hours; p = 0.308, ANCOVA — Group difference (REVAMP - In-person) in mean CPAP daily use over all days adjusted for investigative site; The lower bound of the 95% noninferiority confidence interval was -0.22; Mean Difference (Final Values) = 0.39, Standard Error of Mean 0.37

ADVERSE EVENTS:
Time Frame: Baseline, 1 month and 3 months
Description: Adverse events collected at each scheduled participant encounter and whenever participant contacted research team to report an adverse event.
Arm/Group | REVAMP | In-person Management
All-Cause Mortality (participants affected / at risk) | 0/218 | 0/217
Serious Adverse Events (participants affected / at risk) | 0/218 | 0/217
Other Adverse Events (participants affected / at risk) | 0/218 | 2/217
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | REVAMP (N=218) | In-person Management (N=217)
CPAP mask irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Elective knee surgery (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Not study related

LIMITATIONS AND CAVEATS:
The last participant seen/received an intervention on January 31, 2021.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-20): https://cdn.clinicaltrials.gov/large-docs/45/NCT03007745/Prot_SAP_001.pdf